CLINICAL TRIAL: NCT06207318
Title: Acceptance and Commitment Therapy for the Perioperative Period of Coronary Artery Bypass Graft Surgery: a Randomized Controlled Feasibility Trial
Brief Title: Acceptance and Commitment Therapy for Patients Undergoing Coronary Artery Bypass Graft Surgery
Acronym: ACT for CABG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Sara J. Diesel, Principal Investigator, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202311210
Record Dates: First submitted 2023-12-13; First posted 2024-01-16 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease; Vascularization
Keywords: ACT; CABG
MeSH Terms: conditions — Coronary Artery Disease; Neovascularization, Pathologic | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: The intervention study model will be a two-group, randomized controlled trial. The randomization scheme will follow a 4:1 ratio, with the majority of participants being randomized to the intervention group.
Who Masked: Care Provider
Masking Description: Surgeons, nurses, and other hospital staff involved in patient care will remain blind to psychological treatment condition to avoid potential biases. Laboratory staff processing blood samples for measuring inflammatory biomarkers will be blinded to treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACT Intervention group (Experimental): Participants in the ACT Intervention condition will receive a two-session intervention, with each session lasting 60-90 minutes. Intervention content will center around personal values and behaviors that align with participant goals and utilize the 'triflex' model of ACT, which indicates three core processes of psychological flexibility: be present, open up, and do what matters. Sessions will be facilitated by the PI, an advanced graduate student in the Clinical Science Ph.D. program at the University of Iowa trained in ACT psychotherapy and supervised by a licensed and highly experienced psychologist. Patients will receive a patient workbook and audio recordings of mindfulness exercises that mirror those completed during the session. The intervention will also focus on patients' health-related goals and objectives surrounding their surgery, and expectations for positive post-surgical functioning.
  Interventions: Behavioral: Acceptance and commitment therapy
- Control treatment as usual (TAU) group (No Intervention): The control condition will consist of treatment as usual. This includes a 1.5-hour preoperative appointment with the case-assigned cardiothoracic surgeon and a nurse practitioner. Patients are provided with workbooks that include orientation to the hospital and lifestyle factors information, which includes diet, physical activity, and stress management recommendations.

INTERVENTIONS:
Behavioral: Acceptance and commitment therapy — The intervention will be based on Acceptance and Commitment Therapy (ACT). ACT is an empirically-based therapeutic approach that focuses on psychological flexibility, acceptance, and the reduction of experiential avoidance. It encourages individuals to change their relating to thoughts and experiences and act in accordance with their values.
  Arms: ACT Intervention group

SUMMARY:
Heart disease is the leading cause of death globally, accounting for 16% of the world's total deaths. The number of cases is expected to increase as our population ages. Heart disease also results in large economic burden. It costs the United States about $219 billion per year. Some patients have symptoms that aren't helped by drugs or other medical treatments. These patients will need a surgery that is called cardiac artery bypass graft (CABG) surgery. CABG helps to improve chest pain which is one of the most common complaints of heart disease, and has life-prolonging potential. A limitation of CABG is that it results in increased inflammation. These patients also report high levels of anxiety and depression. Depression and anxiety in the several days surrounding surgery are related to several important things. These include worse health outcomes, worse quality of life, increased risk of death, and increased health care cost. Acceptance and Commitment Therapy (ACT) is a kind of therapy. ACT is adaptable, easy to access, and effective in brief formats. ACT has been gaining evidence for its use in many patient samples. Few studies have used ACT with heart disease patients. No known studies currently exist that have used ACT within the few days surrounding CABG surgery. To address this need, the investigators will conduct a two-arm feasibility randomized control trial (RCT). Patients will be randomized to one of two groups. The first group will complete a brief, 2-session telehealth ACT intervention. The second group will be a control group. The control will consist of treatment as usual. The investigators will evaluate the feasibility of this brief ACT intervention delivered in the peri-operative period. The investigators will also examine preliminary efficacy of the ACT intervention. The investigators will examine anxiety, depression, psychological inflexibility, well-being, and cardiovascular health-related quality of life. The investigators will also examine the intervention's impact on inflammation by measuring two inflammatory markers. The results from this study will also lay the groundwork for larger or multiple site RCT studies.

ELIGIBILITY:
Inclusion Criteria:

* admission to the Heart and Vascular Center at University of Iowa Hospitals and Clinics (UIHC) for urgent or elective CABG
* access to a personal phone or device with video or audio capabilities
* ability to provide informed consent
* English fluency.

Exclusion Criteria:

* life-threatening comorbid (noncardiac) medical condition(s)
* active suicidal ideation or intent
* psychotropic medication use lasting less than four weeks
* inability to provide informed consent and comply with study procedures
* those undergoing repeat revascularization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Theoretical Framework of Acceptability (TFA) questionnaire | 8 weeks
  The TFA is comprised of seven constructs: affective attitude, burden, ethicality, perceived effectiveness, intervention coherence, self-efficacy, and opportunity costs, and also includes an overall acceptability rating. The TFA can be used to generate a single acceptability score and/or to assess the unique domains of acceptability included in the model. Scale scores range from minimum values of 7, and maximum values of 35, with higher scores indicating higher acceptability.
Participant Satisfaction measure | 8 weeks
  Participants will answer five questions on a 5-point Likert-type scale (1 = not at all, 5 = extremely). Scale scores range from minimum values of 5, and maximum values of 25, with higher scores indicating higher satisfaction.
Participant Adherence measure | 8 weeks
  The extent to which participants adhere to the intervention will be assessed via a self-rated measure in which completion of between-session mindfulness and reflection exercises will be reported. Participants will answer four yes/no items. Scale scores range from minimum values of 0, and maximum values of 4, with higher scores indicating higher adherence.
Participant Enrollment | Baseline
  The number and percentage of patients undergoing CABG who are eligible for the study will be tracked as well as the number of participants enrolled in the study. These values will be used to determine the enrollment rate. Additionally, the investigators will track basic patient characteristics such that representativeness of the enrolled sample may be compared to all eligible patients who were approached.
Intervention Delivery | 8 weeks
  Treatment fidelity will be assessed via coder-rated evaluation of interventionist adherence to the manualized treatment protocol. The coder will be a licensed therapist with specific expertise in ACT therapeutic principles and psychotherapy. A randomly selected 20% of sessions will be assessed for treatment fidelity and intervention adherence.
Completion of Study Procedures | 8 weeks
  Completion of all psychological, acceptance, satisfaction, and adherence measures will also be assessed. This will include completion of the entire measure as well as per-item completion which will be recorded for each participant in order to quantify missing data. Attendance will be recorded by the interventionist at each session.
Retention | 8 weeks
  The investigators will assess retention rate by tracking the proportion of enrolled participants who complete all intervention sessions and study procedures.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | 8 weeks
  The PHQ-9 is a self-administered focused measure of depression based on Diagnostic and Statistical Manual of Mental Disorders (DSM) criteria that is utilized for screening, diagnostic, and treatment monitoring purposes. The measure's nine items range from zero (not at all) to three (nearly every day). PHQ-9 scores greater than or equal to five, 10, 15, and 20 out of 27 represent mild, moderate, moderately severe, and severe depression, respectively.
Generalized Anxiety Disorder Questionnaire (GAD-7) | Baseline and 8 weeks
  The Generalized Anxiety Disorder (GAD)-7 survey. The GAD-7 is a self-rated measure designed to screen, measure, and assess the severity of GAD. The seven items range from zero (not at all) to three (nearly every day). Scores greater than or equal to five, 10, and 15 out of 21 represent mild, moderate, and severe anxiety, respectively.
Mental Health Continuum-Short Form (MHC-SF) | Baseline and 8 weeks
  The Mental Health Continuum-Short Form (MHC-SF) is a 14-item scale that is comprised of three subscales: emotional well-being (three items), psychological well-being (six items), and social well-being (five items). Each item measures a distinct dimension of these subscales. The frequency in the past month of each aspect of well-being is rated on a six-point Likert scale (never, once or twice a month, about once a week, two to three times a week, almost every day, every day).
MacNew Heart Disease Health Related Quality of Life (HRQoL) | Baseline and 8 weeks
  The MacNew Heart Disease HRQoL is a self-administered disease-specific questionnaire designed to measure HRQoL in patients with cardiac disease. The measure consists of 27 items that are categorized within three domains: emotional functioning (14 items), physical limitation (13 items), and social functioning (13 items), with 12 items falling into more than one domain. Five items inquire about symptoms such as angina/chest pain, shortness of breath, fatigue, dizziness, and aching legs. The time frame for the MacNew is the previous two weeks. The measure provides both individual scores for each domain as well as a global HRQoL score. Scores range from one (poor HRQoL) to seven (high HRQoL) in each of the three domains.
Comprehensive Assessment of Acceptance Commitment Therapy Processes (CompACT)-15 | Baseline and 8 weeks
  The CompACT-15 assesses psychological inflexibility, experiential avoidance, and maladaptive coping that was adapted to fit the three-factor model of psychological flexibility more adequately and efficiently. This fifteen-item measure utilizes a seven-point Likert scale, ranging from one (strongly disagree) to seven (strongly agree). Scores range from 15 to 105, with higher scores indicating greater psychological flexibility. Three domains are captured within the measure including openness to experience, behavioral awareness, and valued action.
interleukin 6 (IL-6) | Baseline and 8 weeks
  Concentrations of IL-6 will be quantified as indicators of inflammatory processes using a commercially available enzyme-linked immunoassay (ELISA).
high sensitivity c-reactive protein (hs-CRP) | Baseline and 8 weeks
  Concentrations of hs-CRP will be quantified as indicators of inflammatory processes using a commercially available enzyme-linked immunoassay (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Sara J Diesel, MA, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No